CLINICAL TRIAL: NCT07227181
Title: Effects of Animal-Assisted Therapy on Trauma Patient's Willingness to Participate in Ambulation
Brief Title: 2025 Animal Assisted Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Bernard (Other)
Responsible Party: Sponsor-Investigator, Andrew Bernard, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104486
Record Dates: First submitted 2025-11-09; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Trauma; Hospitalized Adult Patients; Rehabilitation; Physical Mobility Impairment; Therapy Dog
Keywords: Animal-Assisted Therapy; Therapy Dog; Trauma Patients; Early Mobilization; Anxiety Reduction; Pain Reduction; Human-Animal Interaction
MeSH Terms: conditions — Anxiety Disorders; Wounds and Injuries; Human-Animal Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Animal-assisted intervention (Experimental): Trauma patients participating in Animal Assisted Intervention
  Interventions: Other: Therapy Dog; Other: Standard mobilization

INTERVENTIONS:
Other: Therapy Dog — Patients assigned to AAI in the morning received standard mobilization in the afternoon, and vice versa. In the AAI intervention, patients interacted with the therapy dog and handler
Other: Standard mobilization — Patients assigned to AAI in the morning received standard mobilization in the afternoon, and vice versa. Standard mobilization no therapy dog is present

SUMMARY:
This study looks at whether walking with a therapy dog helps adult trauma patients move more during their hospital stay. Early movement after an injury or surgery can prevent problems such as blood clots, pressure sores, and muscle loss, but pain and anxiety often make it hard for patients to get out of bed.

Each patient in this study takes part in two walking sessions-one with a certified therapy dog and one without a dog. The order is randomized, so some patients walk with the dog first and others walk without the dog first. Before and after each walk, patients fill out short surveys about their pain, anxiety, and motivation to move. The research team measures how far and how long each patient walks in both sessions.

The goal of this project is to see if therapy dog visits can safely and effectively improve mobility, reduce pain and anxiety, and make walking more enjoyable for trauma patients. Findings from this study may help hospitals design better rehabilitation programs that use animal-assisted therapy to support physical and emotional recovery.

DETAILED DESCRIPTION:
Early mobilization after traumatic injury is a key component of recovery and is associated with reduced complications, shorter hospital stays, and improved functional outcomes. However, trauma patients frequently experience significant barriers to early ambulation, including pain, anxiety, fatigue, and psychological distress following injury and surgery. Animal-assisted interventions (AAI) have demonstrated benefits in reducing pain and anxiety, enhancing mood, and improving patient motivation in various hospital settings. Despite these findings, limited research has examined the role of therapy dogs in promoting early mobility specifically among adult trauma inpatients.

This randomized crossover trial investigates the effect of animal-assisted ambulation on walking duration, distance, and patient-reported outcomes among adult trauma patients admitted to an academic Level I trauma center. Each enrolled participant completes two ambulation sessions within their hospital stay: one with the presence of a certified therapy dog and handler, and one without a dog (standard physical therapy or nursing-led walk). The order of sessions is randomized to control for order effects, and all participants serve as their own control.

During each session, objective ambulation data-including walking duration (minutes), and assistance level-are recorded by the research team or physical therapy staff. Pre- and post-session self-report measures assess pain (DVPRS), anxiety (Modified GAD-7), and motivation to mobilize (Likert scale).

The study aims to evaluate whether therapy dog-assisted ambulation results in greater walking duration and distance, as well as reduced perceived pain and anxiety, compared to standard ambulation without a therapy dog. Secondary analyses will explore potential moderating effects of time of day, patient demographics, and mechanism of injury on intervention effectiveness.

All therapy dogs and handlers are registered through a national certification organization and follow strict infection control and safety protocols consistent with institutional policy. Data will be analyzed using mixed-effects models to account for within-subject correlations and to assess crossover effects.

This study is designed to inform evidence-based integration of animal-assisted therapy into trauma rehabilitation protocols, supporting both the physical and psychosocial dimensions of recovery in hospitalized trauma patients

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age and older)
* trauma patients

Exclusion Criteria:

* weight bearing limitation
* spine instability
* oxygen requirement >2LPM, GCS <15,
* high fall risk (as evidenced by door label)
* fear of dogs
* allergies to dogs
* prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-23 (Actual)

PRIMARY OUTCOMES:
Change in Defense & Veterans Pain Rating Scale | baseline and post intervention (1 day)
  Before and after each intervention, patients completed surveys assessing pain using the (Defense and Veterans Pain Rating Scale, DVPRS). Scores on the scale ranged from 0: no pain to 10: worst pain of patient's life.
Change in General Anxiety Disorder-7 (GAD-7) Scale | Baseline and post intervention (1 day)
  Before and after each intervention, patients completed surveys assessing anxiety using modified General Anxiety Disorder-7 (GAD-7). Scaled from not at all to a lot, resulting in a total score that can range from 0 to 21, with higher values reflecting more severe anxiety symptoms.
General status | baseline and post intervention (1 day)
  Before and after each intervention, patients completed surveys assessing general status. Used likert scale ranging from very poor to excellent.
Willingness to mobilize | baseline and post intervention (1day)
  Before and after each intervention, patients completed surveys assessing willingness to mobilize. Used likert scale ranging from no motivation at all to very much.
Mobilization difficulty | Baseline and post intervention (1 day)
  Before and after each intervention, patients completed surveys assessing mobilization difficulty. Used likert scale ranging from very easy to very hard.
Overall mobility satisfaction | Baseline and post intervention (1 day)
  Before and after each intervention, patients completed surveys assessing overall mobility satisfaction. Used likert scale ranging from not satisfied to very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bernard, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Albert B. Chandler Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No